CLINICAL TRIAL: NCT00725153
Title: Evaluation of Deposits on Contact Lenses Worn Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MS-006
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-07

CONDITIONS: Refractive Error
Keywords: Contact lens deposits; Soft contact lenses; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PureVision/Acuvue 2 (Other): PureVision contact lenses worn first, with Acuvue 2 contact lenses worn second. Both products worn for 10 hours each.
  Interventions: Device: Balafilcon A contact lenses (PureVision); Device: Etafilcon A contact lenses (Acuvue2)
- Acuvue 2/PureVision (Other): Acuvue 2 contact lenses worn first, with PureVision contact lenses worn second. Both products worn for 10 hours each.
  Interventions: Device: Balafilcon A contact lenses (PureVision); Device: Etafilcon A contact lenses (Acuvue2)

INTERVENTIONS:
Device: Balafilcon A contact lenses (PureVision) — Commercially marketed, soft contact lenses worn bilaterally for 10 hours
  Other Names: PureVision
Device: Etafilcon A contact lenses (Acuvue2) — Commercially marketed, soft contact lenses worn bilaterally for 10 hours
  Other Names: Acuvue2

SUMMARY:
The purpose of this study was to measure front surface deposits on contact lenses when worn for ten hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Visual acuity correctable to 20/30 (Snellen) or better in each eye at distance with contact lenses.
* Successfully wearing hydrogel or silicone hydrogel contact lenses prior to enrollment in the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Evidence or history of keratitis (dendritic keratitis); viral disease of the cornea and/or conjunctiva; acute bacterial disease of the cornea and/or conjunctiva and/or eyelids; infection of the eye; and/or fungal disease of the eye.
* One functional eye or a monofit lens.
* Ocular conditions such as active acute blepharitis, conjunctival infections, and iritis.
* Any slit-lamp finding score of (1) at the Screening Visit as defined in protocol.
* Use of concomitant topical ocular prescription or over-the-counter (OTC) ocular medications.
* History of seasonal allergies with significant ocular side effects which may have an adverse impact on contact lens wear.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 Subjects currently wearing hydrogel or silicone hydrogel lenses were recruited at 3 US and 1 United Kingdom study sites.
Pre-assignment Details: Subjects randomized by lens order to wear PureVision and Acuvue 2 lenses for 10 hours each.
Groups:
- PureVision / Acuvue 2: PureVision lenses worn in Period One, Acuvue 2 lenses worn in Period Two. Both products worn for 10 hours each.
- Acuvue 2 / PureVision: Acuvue 2 lenses worn in Period One, PureVision lenses worn in Period Two. Both products worn for 10 hours each.
Period: Period One, 10 Hours of Wear
Arm/Group | PureVision / Acuvue 2 | Acuvue 2 / PureVision
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0
Period: Period Two, 10 Hours of Wear
Arm/Group | PureVision / Acuvue 2 | Acuvue 2 / PureVision
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All enrolled participants
Arm/Group | Overall
Number analyzed (Participants) | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 31.95 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Front Surface Lens Deposits
Description: Film and discrete deposits were assessed with a slit-lamp after 10 hours of lens wear. Film deposits were recorded on a 5-point scale, where 0=no deposition, clean surface; 1=slight, deposition occupying 1-5% of lens front surface; 2=mild, deposition occupying 6-15% of lens front surface; 3=moderate, deposition occupying 16-25% of lens front surface; 4=severe, deposition occupying >25% of lens front surface. Discrete deposits were recorded on a 5-point scale, where 0=no deposition, clean surface; 1=microdeposits (less than or equal to 10 dots); 2=microdeposits (greater than 10 dots); 3=macro deposits; 4=one or more jelly bumps. Participants were classified into Front Surface Lens Deposits <2 (less than grade 2 for both film and discrete) and into front surface lens deposits >1 (greater than grade 1 for either film, discrete, or both).
Time Frame: 10 hours
Population: All enrolled participants.
Measure: Number; unit: Participants
Groups:
- PureVision Contact Lenses: PureVision lenses worn 10 hours
- Acuvue 2 Contact Lenses: Acuvue 2 lenses worn 10 hours
Arm/Group | PureVision Contact Lenses | Acuvue 2 Contact Lenses
Number analyzed (Participants) | 55 | 55
Participants
  Deposits Graded <2 | 27 | 32
  Deposits Graded >1 | 28 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: Safety data was collected on all enrolled and dispensed subjects.
Groups:
- PureVision Lenses Worn 10 Hours: PureVision lenses worn 10 hours
- Acuvue 2 Lenses Worn 10 Hours: Acuvue 2 lenses worn 10 hours
Arm/Group | PureVision Lenses Worn 10 Hours | Acuvue 2 Lenses Worn 10 Hours
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less